CLINICAL TRIAL: NCT02666209
Title: Early Patient Access Single Named Patient Program for the Use of Ulocuplumab for the Treatment of Multiple Myeloma
Status: No longer available | Type: Expanded Access
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Irene Ghobrial, MD, Irene M. Ghobrial, MD, Dana-Farber Cancer Institute
Other Study IDs: 16-002; CA212-122 (Other: Bristol-Myers Squibb)
Record Dates: First submitted 2016-01-22; First posted 2016-01-28 (Estimated); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: Multiple Myeloma in Relapse; Multiple Myeloma
Keywords: Multiple Myeloma; Relapsed Multiple Myeloma; Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — ulocuplumab; Lenalidomide; Bortezomib; Dexamethasone; Calcium Dobesilate

INTERVENTIONS:
Drug: Ulocuplumab — CXCR4 inhibitor given weekly on a 28 day cycle intravenously
  Other Names: BMS-936564
Drug: Lenalidomide — immunomodulatory agent given days 1-21 of a 28 day cycle orally in subjects not receiving bortezomib
  Other Names: Revlimid
Drug: Bortezomib — proteasome inhibitor given at physician discretion in subjects not receiving lenalidomide
  Other Names: Velcade
Drug: Dexamethasone — steroid given at physician discretion on a 28 day cycles
  Other Names: Decadron

SUMMARY:
Participant that has been diagnosed with Relapsed/ Refractory Multiple Myeloma and are currently participating in a clinical trial which is closing. This research study is studying Ulocuplumab as a possible treatment. It's an expanded access from NCT01359657

DETAILED DESCRIPTION:
This research study is an Expanded Access Trial, which is a way to provide an investigational therapy to individuals who are not eligible to receive that therapy in a clinical trial, but have a serious or life-threatening illness for which other treatments are not available.

The purpose of this expanded access program is to treat participants diagnosed with relapsed or refractory multiple myeloma with an investigational drug called ulocuplumab.

Participants enrolled in the program will receive ulocuplumab with lenalidomide and dexamethasone or ulocuplumab with bortezomib and dexamethasone. Ulocuplumab is supposed to kill myeloma cells.

Lenalidomide, which is also known as Revlimid® and Bortezomib, which is also known as Velcade®, are approved by the FDA for treatment of Multiple Myeloma. Dexamethasone, also known as Decadron®, is also approved by the FDA for other treatments. It is a type of steroid medication that fights inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent document
* Must be currently participating on protocol 11-240 (DFCI)/ CA 212-002(BMS), tolerating therapy, and still receiving benefit from treatment.

Exclusion Criteria:

* Prior exposure to Ulocuplumab other than in DFCI Protocol 11-240 (BMS protocol CA212-002) or any other any other CXCR4 inhibitor (small molecule within 14 days; antibody against CXCR4 within 10 weeks).

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Irene M Ghobrial, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States